CLINICAL TRIAL: NCT03040466
Title: Randomized Controlled Trial Comparing Disposable to Reusable Flexible Ureteroscope for Treatment of Upper Urinary Tract Stone
Brief Title: Comparing Treatment of Urolithiasis Between Disposable and Reusable Ureteroscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-20844
Record Dates: First submitted 2017-01-23; First posted 2017-02-02 (Estimated); Results first posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Kidney Calculi; Ureter Calculi
Keywords: ureteroscopy; flexible ureteroscope; randomized controlled trial
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to each 3 type of ureteroscope and receive the flexible ureteroscopy. In each ureteroscopy, only one type of ureteroscope will be used; therefore this study will be parallel model.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- reusable fiberoptic ureteroscope (Active Comparator): For this arm, participants will receive the ureteroscopy for their kidney and ureter stones using reusable fiberoptic flexible ureteroscope (URF-P6, Olympus). The surgical method of the ureteroscopy will be a standard fashion same as other arms.
  Interventions: Device: reusable fiberoptic ureteroscope
- disposable digital ureteroscope (Experimental): For this arm, participants will receive the ureteroscopy for their kidney and ureter stones using disposable digital flexible ureteroscope (LithoVue, Boston Scientific). The surgical method of the ureteroscopy will be a standard fashion same as other arms.
  Interventions: Device: disposable digital ureteroscope

INTERVENTIONS:
Device: reusable fiberoptic ureteroscope — We will use reusable fiberoptic ureteroscopes for the treatment of kidney and ureter stones.
  Arms: reusable fiberoptic ureteroscope
Device: disposable digital ureteroscope — We will use disposable digital ureteroscopes for the treatment of kidney and ureter stones.
  Arms: disposable digital ureteroscope

SUMMARY:
Reusable flexible ureteroscopes are widely used to treat various upper urinary tract diseases including urinary stones. However, they require a long turnover time between procedures because of the sterilization process. Moreover, repeated use of a scope ultimately deteriorates its image quality which leads to a high maintenance cost in the long-term. A disposable digital flexible ureteroscope was released in the United States in January 2016, offering an improved image resolution, new scope performance characteristics with every case, and no need for sterilization and repair. Preliminary data from our center has demonstrated that disposable scopes shorten operative time by 25% compared to reusable fiberoptic scope and are associated with a 2/3 reduction in procedural complication rate. Therefore, treatment with disposable scopes may be more effective for patients and facilitate cost management within the hospital.

Here, we propose a three-armed, prospective randomized study, comparing treatment outcomes between disposable digital, reusable fiberoptic, and reusable digital flexible ureteroscopes.

DETAILED DESCRIPTION:
This is a single center, prospective, randomized controlled pragmatic clinical trial designed to compare between disposable, reusable fiberoptic, and reusable digital ureteroscopes in upper urinary tract stone treatment efficacy. Three hundred subjects with kidney and/or ureteral stones are planned to recruit for the study. All subjects will be computer sequence-randomized into having their ureteroscopic treatment performed with a disposable (LithoVue™), reusable fiberoptic (URF-P6™), or reusable digital (URF-V2™) flexible ureteroscope. Patient's demographics, physical, laboratory, and image findings will be collected before surgery. These clinical data are already being collected as part of an ongoing registry study. Perioperative timing as well as operator's satisfaction and fatigue and need for a second ureteroscope during the case will be recorded during the treatment course. Other clinical data will be collected at days 7, 30, 90, 180 after surgery. The condition of the used ureteroscopes will be tracked and recorded to confirm the repair rate.

Screening data will be reviewed to determine subject eligibility. Subjects who meet all inclusion criteria and none of the exclusion criteria will be entered into the study.

The following surgical treatment will be used similarly for all three randomized arms and represents standard of case therapy:

Ureteroscopic stone removal Under general anesthesia, the patient is placed in the lithotomy position. All procedures are performed under direct videoscopic and fluoroscopic guidance. Fluoroscopic screening is utilized using a mobile multidirectional C-arm fluoroscopy unit. Initially, a safety guide-wire is placed into the renal pelvis, followed by a ureteral access sheath as needed to maintain low intra-renal pressure and to facilitate the procedures. Using a flexible ureteroscope, renal or ureteral stones are identified and fragmented with a holmium YAG laser. Basket extraction of residual fragments is done until visual complete clearance of stone fragments is achieved.

After ureteroscopy is done and stone clearance is achieved, a ureteral stent is placed at the end of the procedure to drain the kidney for 2-21 days if it is clinically indicated.

The total duration of the study is expected to be one year for subject recruitment and one year and six months for final subject follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age at their first clinical visit.
2. Patients with either unilateral or bilateral upper urinary tract stone of any size and location, treatable by flexible ureteroscopy, diagnosed by preoperative ultrasound, computed tomography or plain radiographic imaging
3. Patients being able and willing to provide consent.

Exclusion Criteria:

1. Serious illness likely to cause death within the next 5 years, so as to exclude significant metabolic derangements that might lead to adverse surgical outcome.
2. Pregnancy.
3. Staged ureteroscopic procedure.
4. Antegrade flexible ureteroscopy.
5. Dual procedures (ureteroscopy concurrently performed with other operations).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Chi, MD, Principal Investigator — Urology, University of California San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Healy KA, Pak RW, Cleary RC, Colon-Herdman A, Bagley DH. Hand problems among endourologists. J Endourol. 2011 Dec;25(12):1915-20. doi: 10.1089/end.2011.0128. Epub 2011 Oct 17. PMID 22004843
- [Background] Karaolides T, Bach C, Kachrilas S, Goyal A, Masood J, Buchholz N. Improving the durability of digital flexible ureteroscopes. Urology. 2013 Apr;81(4):717-22. doi: 10.1016/j.urology.2013.01.016. Epub 2013 Mar 7. PMID 23465156
- [Background] Multescu R, Geavlete B, Geavlete P. A new era: performance and limitations of the latest models of flexible ureteroscopes. Urology. 2013 Dec;82(6):1236-9. doi: 10.1016/j.urology.2013.07.022. Epub 2013 Aug 28. PMID 23992972
- [Background] Somani BK, Al-Qahtani SM, de Medina SD, Traxer O. Outcomes of flexible ureterorenoscopy and laser fragmentation for renal stones: comparison between digital and conventional ureteroscope. Urology. 2013 Nov;82(5):1017-9. doi: 10.1016/j.urology.2013.07.017. Epub 2013 Aug 31. PMID 24001703
- [Background] Carey RI, Martin CJ, Knego JR. Prospective evaluation of refurbished flexible ureteroscope durability seen in a large public tertiary care center with multiple surgeons. Urology. 2014 Jul;84(1):42-5. doi: 10.1016/j.urology.2014.01.022. Epub 2014 May 14. PMID 24837456
- [Background] de la Rosette J, Denstedt J, Geavlete P, Keeley F, Matsuda T, Pearle M, Preminger G, Traxer O; CROES URS Study Group. The clinical research office of the endourological society ureteroscopy global study: indications, complications, and outcomes in 11,885 patients. J Endourol. 2014 Feb;28(2):131-9. doi: 10.1089/end.2013.0436. Epub 2013 Dec 17. PMID 24147820
- [Background] Geavlete P, Multescu R, Geavlete B. Pushing the boundaries of ureteroscopy: current status and future perspectives. Nat Rev Urol. 2014 Jul;11(7):373-82. doi: 10.1038/nrurol.2014.118. Epub 2014 Jun 3. PMID 24890883
- [Background] Tosoian JJ, Ludwig W, Sopko N, Mullins JK, Matlaga BR. The effect of repair costs on the profitability of a ureteroscopy program. J Endourol. 2015 Apr;29(4):406-9. doi: 10.1089/end.2014.0435. Epub 2014 Nov 7. PMID 25286008
- [Background] Buttice S, Sener TE, Netsch C, Emiliani E, Pappalardo R, Magno C. LithoVue: A new single-use digital flexible ureteroscope. Cent European J Urol. 2016;69(3):302-305. doi: 10.5173/ceju.2016.872. Epub 2016 Aug 26. No abstract available. PMID 27730000
- [Background] Doizi S, Kamphuis G, Giusti G, Andreassen KH, Knoll T, Osther PJ, Scoffone C, Perez-Fentes D, Proietti S, Wiseman O, de la Rosette J, Traxer O. First clinical evaluation of a new single-use flexible ureteroscope (LithoVue): a European prospective multicentric feasibility study. World J Urol. 2017 May;35(5):809-818. doi: 10.1007/s00345-016-1936-x. Epub 2016 Sep 26. PMID 27671898
- [Background] Martin CJ, McAdams SB, Abdul-Muhsin H, Lim VM, Nunez-Nateras R, Tyson MD, Humphreys MR. The Economic Implications of a Reusable Flexible Digital Ureteroscope: A Cost-Benefit Analysis. J Urol. 2017 Mar;197(3 Pt 1):730-735. doi: 10.1016/j.juro.2016.09.085. Epub 2016 Sep 28. PMID 27693449
- [Result] Usawachintachit M, Isaacson DS, Taguchi K, Tzou DT, Hsi RS, Sherer BA, Stoller ML, Chi T. A Prospective Case-Control Study Comparing LithoVue, a Single-Use, Flexible Disposable Ureteroscope, with Flexible, Reusable Fiber-Optic Ureteroscopes. J Endourol. 2017 May;31(5):468-475. doi: 10.1089/end.2017.0027. Epub 2017 Mar 13. PMID 28287823

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Reusable Fiberoptic Ureteroscope | Disposable Digital Ureteroscope
Started | 65 | 115
Completed | 65 | 115
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reusable Fiberoptic Ureteroscope | Disposable Digital Ureteroscope | Total
Number analyzed (Participants) | 65 | 115 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (12.6) | 55.8 (15.1) | 53.8 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 54 | 88
  Male | 31 | 61 | 92
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 65 | 115 | 180

OUTCOME MEASURES:

1. Primary Outcome: Overall Procedure Time
Time Frame: at the surgery day, this will be a duration that each ureteroscopy is performed for a patient, assessed between 10 and 120 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Reusable Fiberoptic Ureteroscope | Disposable Digital Ureteroscope
Number analyzed (Participants) | 65 | 115
minutes | 64.5 (37.0) | 54.1 (25.7)

2. Secondary Outcome: Number of Participants That Are Stone Free
Description: this will be determined by either CT, US, or KUB
Time Frame: three month after surgery
Population: Postoperative imaging was requested of all patients, but the total study group did not follow up with kidney, ureter, and bladder radiograph or ultrasound surveillance imaging. Participants with post operative imaging included here.
Measure: Count of Participants; unit: Participants
Arm/Group | Reusable Fiberoptic Ureteroscope | Disposable Digital Ureteroscope
Number analyzed (Participants) | 38 | 40
Participants | 17 | 24

3. Secondary Outcome: Number of Participants With Complications
Time Frame: from during the surgery to three months after the surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Reusable Fiberoptic Ureteroscope | Disposable Digital Ureteroscope
Number analyzed (Participants) | 65 | 115
Participants | 9 | 9

ADVERSE EVENTS:
Arm/Group | Reusable Fiberoptic Ureteroscope | Disposable Digital Ureteroscope
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/115
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/115
Other Adverse Events (participants affected / at risk) | 9/65 | 9/115
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Reusable Fiberoptic Ureteroscope (N=65) | Disposable Digital Ureteroscope (N=115)
Presence of postoperative complications (Surgical and medical procedures) | 9 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No